CLINICAL TRIAL: NCT02518035
Title: Use of Silicone Gel to Improve Retroauricular Scar in Microtia Patients
Brief Title: Silicone Gel to Improve Scar in Microtia Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 103-2849B
Record Dates: First submitted 2015-08-05; First posted 2015-08-07 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-07

CONDITIONS: Microtia; Scar
MeSH Terms: conditions — Congenital Microtia; Cicatrix | interventions — Silicone Gels

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Placebo Comparator): No silicone gel treatment after remove of stitches
- Experimental (Experimental): Silicone gel applied for twice per day
  Interventions: Drug: Silicone Gel

INTERVENTIONS:
Drug: Silicone Gel — Silicone gel will be applied twice per day in the experimental group
  Other Names: Dermatix Ultra Gel
  Arms: Experimental

SUMMARY:
Effort to reduce post-surgical scar is especially important for microtia patients. Even the scar lies posterior to ear auricle, but hypertrophic scar contracture may limit the ear auricle projection. If the scar is hypertrophic and conspicuous, this stigmata will accompanies the child for many years.The main objective aim of this study is to examine whether post-operative use of silicone gel can improve scar formation for microtia reconstruction scars.

DETAILED DESCRIPTION:
Background:

A scar represents dermal fibrous replacement tissue and results from a wound that has healed by resolution rather than regeneration. Undesirable scars, such as hypertrophic or keloid scars, occur most frequently over the anterior chest, shoulders, scapular area, lower abdomen and suprapubic region. Many of the investigators' microtia patients complained postsurgical hypertrophic scar. The incidence of hypertrophic scars after microtia reconstruction could be 6.29%.

Effort to reduce post-surgical scar is especially important for microtia patients. Even the scar lies posterior to ear auricle, but hypertrophic scar contracture may limit the ear auricle projection. If the scar is hypertrophic and conspicuous, this stigmata will accompanies the child for many years. The micropore tapes is very useful for facial scars. However, because of retroauricular contour and hairline, micropore tapes is difficult to retained over it place. Self-dry silicone gel is effective in both treatment and prevention of hypertrophic scar. It is consider first line for hypertrophic prevention in last update of facial scar care.

The main objective aim of this study is to examine whether post-operative use of silicone gel can improve scar formation for microtia reconstruction scars.

Patients and Methods:

This is a prospective randomize clinical trial primarily designed to compare the scarring after second stage of microtia repair with post-operative use of self-drying silicone gel. The control group did not use self-drying silicone gel for their scar care. The study group will receive application of self-dry silicone gel (Dermatix Ultra Gel - Invida, Hanson Medical Inc, USA) twice a day.

Six months after surgery, Vancouver scar sale and Visual analogue scale will be used for subjective scar measurement. Standard craniofacial photograph will be taken at the same time. A surgical ruler will be placed underneath the op wound. The scar width will be measured using with commercial software.

ELIGIBILITY:
Inclusion Criteria:

* Patients with microtia.
* Written informed consent given by parent/guardian.

Exclusion Criteria:

* Combined other craniofacial anomalies
* Without permission of parent/guardian, without signed informed consent by parent/guardian.

Ages: 9 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Scar width | 6 months after surgery
  6 months after surgery, the scar width will be measured

SECONDARY OUTCOMES:
Vancouver Scar Scale | 6 months after surgery
  6 months after surgery, the scar quality will be assessed with Vancouver Scar
Visual Analogue Scale | 6 months after surgery
  6 months after surgery, the scar will be assessed with visual analogue scale of 10 grade

CONTACTS AND LOCATIONS:
Overall Officials: Zung-Chung Chen, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Chun Shin, Taoyuan District, Taiwan

REFERENCES:
- [Background] Chen ZC, Chen K, Jo LJ, Nagata S. Satisfactory reconstruction with autologous costal cartilage graft in a geriatric microtia patient. Plast Reconstr Surg. 2009 Jan;123(1):1e-6e. doi: 10.1097/PRS.0b013e3181934660. No abstract available. PMID 19116506
- [Background] Chen ZC, Chen PK, Hung KF, Lo LJ, Chen YR. Microtia reconstruction with adjuvant 3-dimensional template model. Ann Plast Surg. 2004 Sep;53(3):282-7. doi: 10.1097/01.sap.0000106434.69246.29. PMID 15480018
- [Background] Chen ZC, Goh RCW, Chen PK, Lo LJ, Wang SY, Nagata S. A new method for the second-stage auricular projection of the Nagata method: ultra-delicate split-thickness skin graft in continuity with full-thickness skin. Plast Reconstr Surg. 2009 Nov;124(5):1477-1485. doi: 10.1097/PRS.0b013e3181babaf9. PMID 20009834
- [Background] Chen ZC, Albdour MN, Lizardo JA, Chen YA, Chen PK. Precision of three-dimensional stereo-photogrammetry (3dMD) in anthropometry of the auricle and its application in microtia reconstruction. J Plast Reconstr Aesthet Surg. 2015 May;68(5):622-31. doi: 10.1016/j.bjps.2015.02.020. Epub 2015 Mar 9. PMID 25892285
- [Background] Wallace CG, Mao HY, Wang CJ, Chen YA, Chen PK, Chen ZC. Three-dimensional computed tomography reveals different donor-site deformities in adult and growing microtia patients despite total subperichondrial costal cartilage harvest and donor-site reconstruction. Plast Reconstr Surg. 2014 Mar;133(3):640-651. doi: 10.1097/01.prs.0000438052.14011.0a. PMID 24572854